CLINICAL TRIAL: NCT03660488
Title: Clinical Trial Evaluating the Clinical Efficacy of Cefixime for Treatment of Early Syphilis
Brief Title: Cefixime for Alternative Syphilis Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: AIDS Healthcare Foundation (Other)
Responsible Party: Principal Investigator, Jeffrey D. Klausner, MD, MPH, Professor of Medicine & Public Health, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-000665; 20181796 (Other: Western IRB)
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Syphilis; Early Syphilis
Keywords: syphilis; cefixime; penicillin
MeSH Terms: conditions — Syphilis | interventions — Cefixime; Penicillin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Benzathine Penicillin G (Active Comparator): Patients of the "Penicillin Group" will receive the standard of care treatment. This is one intramuscular injection of 2.4 million units Benzathine Penicillin G. The group will consist of 50 patients.
  Interventions: Drug: Benzathine Penicillin G
- Cefixime Group (Experimental): Patients of the "Cefixime Group" will receive Cefixime 400 mg, per os, one tablet, two times per day, for ten consecutive days. The study team will provide the medication.
  The group will consist of 50 patients.
  Interventions: Drug: Cefixime 400 milligram Oral Capsule [Suprax]

INTERVENTIONS:
Drug: Cefixime 400 milligram Oral Capsule [Suprax] — The intervention group will receive Cefixime 400mg, one tablet twice per day, for ten consecutive days
  Other Names: Suprax
  Arms: Cefixime Group
Drug: Benzathine Penicillin G — The control group will receive Benzathine Penicillin G 2.4 Million Units intramuscularly for treatment of syphilis. Penicillin is the indicated treatment for syphilis infection
  Arms: Benzathine Penicillin G

SUMMARY:
The goal of the study is to evaluate the efficacy of oral cefixime as an alternative treatment for syphilis infection.

One hundred adult patients (≥18 years old) with syphilis infection (positive Treponema Pallidum Particle Agglutination assay and RPR titer ≥ 1/8) will be recruited. Participants will be randomized (1:1) to receive either the standard of care Penicillin or Cefixime.

During the study, participants will visit the clinic up to 5 times; at baseline visit, at 3, 6, 12 months after treatment initiation. Participants of the cefixime group will be required to visit the clinic 14 days after treatment initiation. In each visit, participants will be asked about current symptoms and do laboratory tests for syphilis (RPR). Subjects who have a 4-fold decrease (from study entry RPR) in RPR titers from baseline at 6 months will be considered a positive treatment response.

DETAILED DESCRIPTION:
Syphilis is a major issue worldwide causing 5.6 million new cases of syphilis worldwide, of which over 900,000 are pregnant women. It is also responsible for congenital infections causing fetal loss or stillbirth or, in a live-born infant, neonatal death, prematurity and low birth weight. Penicillin is the currently used treatment. However, lack of penicillin and alternatives to treatment often hinder treatment and prevention efforts.

Cefixime is an FDA-approved, orally administered third-generation cephalosporin that is currently used for the treatment of a wide range of infections, including urinary tract infections. Our goal is to evaluate the efficacy and safety of oral cefixime as an alternative treatment for syphilis infection.

One hundred adult patients (≥18 years old) with syphilis infection will be recruited. Eligible participants will have laboratory-confirmed syphilis infection with a positive Treponema pallidum Particle Agglutination (TPPA) assay and RPR (Rapid Plasma Reagin ) titer ≥ 1/8. Participants will be randomized (1:1) to receive either the standard of care Penicillin or Cefixime.

During the study, participants will visit the clinic 5 times; at baseline visit, demographic, clinical information and laboratory test results for syphilis will be recorded and treatment will start. Depending on the study group, the treatment plan will be oral Cefixime 400mg, twice per day for ten consecutive days or one dose of intramuscular Penicillin. Patients will be required to visit the clinic two weeks after treatment initiation to verify adverse effects. Follow up visits will occur at 3, 6 and 12 months after treatment initiation. In each visit, participants will be asked about current symptoms, interval sexual history, concomitant antibiotic use and possible adverse reactions. Subjects will also have a venipuncture blood specimen collected for syphilis testing (RPR). Subjects who have a 4-fold decrease (from study entry RPR) in RPR titers from baseline at 6 months will be considered a positive treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older and able to provide informed consent
2. Cases of primary, secondary or early latent syphilis with RPR titer ≥1:8 within 3 weeks prior to enrollment.
3. HIV infected individuals willing to participate in the study must have CD4 count ≥350 cells/μl within the last 4 weeks and be virally suppressed (i.e., viral load ≤ 200 copies/mL) for HIV for the 6 months prior to enrolment with the most recent results within the last 4 weeks. inclusion
4. Non-cephalosporin allergic
5. Able to travel to the clinic once a day or be available for phone calls or receive text messages for at least 7-10 days and willing to attend follow-up visits
6. Able to swallow pills

Exclusion Criteria:

1. Pregnancy or positive pregnancy test
2. Serofast RPR titer (prior titer 1:8 or greater)
3. Recent (less than 7 days) or concomitant antimicrobial therapy with activity against syphilis.
4. Cephalosporin allergy: previous episode of flushing, urticaria, angioedema, rhinitis, bronchospasm, and anaphylactic shock, rash after taking cephalosporin.
5. Penicillin allergy: previous episode of flushing, urticaria, angioedema, rhinitis, bronchospasm, and anaphylactic shock, rash after receiving Penicillin.
6. Has a medical condition or other factor that might affect their ability to follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Klausner, MD MPH, Principal Investigator — University of California, Los Angeles; David Tellalian, MD, Principal Investigator — AIDS Helthcare Foundation
Locations (10):
- United States (10):
  - AHF Westside, Beverly Hills, California
  - AHF Downtown Healthcare Center, Los Angeles, California
  - AHF Carl Bean, Los Angeles, California
  - AHF Hollywood Healthcare Center, Los Angeles, California
  - AHF Wellness on Western Center, Los Angeles, California
  - AHF Oakland Wellness Center, Oakland, California
  - AHF Healthcare Center Oakland, Oakland, California
  - AHF San Francisco, San Francisco, California
  - AHF Valley, Sherman Oaks, California
  - AHF Las Vegas Healthcare Center, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data, participant data will not be provided or shared with other researchers, apart from the members of the research team or regulatory authorities

REFERENCES:
- [Derived] Mehta SN, Stafylis C, Tellalian DM, Burian PL, Okada CM, Millner CE, Mejia CM, Klausner JD. Clinical trial protocol to evaluate the efficacy of cefixime in the treatment of early syphilis. Trials. 2020 Dec 9;21(1):1009. doi: 10.1186/s13063-020-04885-z. PMID 33298143

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefixime Group: Patients of the "Cefixime Group" will receive Cefixime 400 mg, per os, one tablet, two times per day, for ten consecutive days. The study team will provide the medication.
  The group will consist of 50 patients.
  Cefixime 400 milligram Oral Capsule [Suprax]: The intervention group will receive Cefixime 400mg, one tablet twice per day, for ten consecutive days
Period: Overall Study
Arm/Group | Benzathine Penicillin G | Cefixime Group
Started | 31 | 27
Completed | 31 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benzathine Penicillin G | Cefixime Group | Total
Number analyzed (Participants) | 31 | 27 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 26 | 57
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [35.5 to 50.5] | 39 [31.5 to 49] | 39 [36 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 31 | 27 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 37
  Not Hispanic or Latino | 12 | 9 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Hispanic/Latinx, or Spanish Origin | 19 | 18 | 37
  Race/ethnicity: Non-Hispanic African American | 5 | 4 | 9
  Race/ethnicity: Non-Hispanic White | 6 | 4 | 10
  Race/ethnicity: Non-Hispanic Asian/Hawaiian/Pacific Islander | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 27 | 58

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: subjects who have a 4-fold decrease (from study entry Rapid plasma reagin) in Rapid plasma reagintiters from baseline at 3 or 6 months will be considered a positive treatment response.
Time Frame: 3 or 6 months after treatment completion
Measure: Count of Participants; unit: Participants
Arm/Group | Benzathine Penicillin G | Cefixime Group
Number analyzed (Participants) | 15 | 15
Participants | 14 | 13

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the duration of the study (12 months) starting from enrollment. Evaluation for adverse events occurred during follow ups; for the cefixime group we evaluated adverse events during the 10-day visit. Participants and study clinicians were instructed to report any occurrence to the study team for review.
Description: In case of an adverse event, participants were instructed to contact the study team. The team had provided necessary clinic and study team contact informaion
Arm/Group | Benzathine Penicillin G | Cefixime Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/27
Other Adverse Events (participants affected / at risk) | 0/31 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benzathine Penicillin G (N=31) | Cefixime Group (N=27)
Mild Skin Rash (Skin and subcutaneous tissue disorders) | NA | 1 (1) — Skin rash within 24 hours after receiving cefixime

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT03660488/Prot_SAP_001.pdf